CLINICAL TRIAL: NCT06832813
Title: Long Term Efficacy and Safety of Transcranial Magnetic Stimulation Targeting Cerebellum to Treat Drug-resistant Epilepsy During Enhanced and Maintenance Phase
Brief Title: Long Term Efficacy and Safety of TMS Targeting Cerebellum to Treat DRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20252042
Record Dates: First submitted 2025-02-04; First posted 2025-02-18 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-02

CONDITIONS: Drug-resistant Epilepsy; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participant Group (Experimental): Continuous θ-burst stimulation (cTBS) is characterized by plexus stimulation. The stimulation intensity was 80% resting motor threshold (RMT) at 50Hz of intra plexus pulse while the frequency of inter plexus pulse is 5Hz, the duration was 40s, and the number of stimulation pulses was 600. Two groups of stimulation were repeated in each cerebellar dentate nucleus with an interval of 5 min in each group.
  Interventions: Device: cTBS

INTERVENTIONS:
Device: cTBS — Continuous θ-burst stimulation (cTBS) is characterized by plexus stimulation. The stimulation intensity was 80% resting motor threshold (RMT) at 50Hz of intra plexus pulse while the frequency of inter plexus pulse is 5Hz, the duration was 40s, and the number of stimulation pulses was 600. Two groups of stimulation were repeated in each cerebellar dentate nucleus with an interval of 5 min in each group.
  1. Enhanced phase：participants received cTBS treatment for a total of 5 times a week for 2 weeks；
  2. Consolidation phase：participants received cTBS treatment for a total of twice a week (at least 24 hours apart) for 8 weeks；
  3. Maintenance phase：participants received cTBS treatment for a total of once a week for 8 weeks.

SUMMARY:
This study aims to observe the long term efficacy and safety of cerebellar continuous θ burst stimulation (cTBS) for drug-resistant Epilepsy during enhanced and maintenance phase，in order to provide a new treatment for long-term control of drug-resistant epilepsy and improve the quality of life of those patients. A total of 100 patients with DRE will undergo cTBS treatment by precise navigation to bilateral cerebellar dentate nuclei. The frequency and clinical feature of seizures, scalp EEG，clinical score, MOCA，MMSE，and QOLIE-31 were ssessed at baseline, after 2 weeks of enhanced phase，8 weeks of consolidate phase, and 8 weeks of maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old，
2. Participants who are diagnosed as drug- resistant epilepsy,
3. Participants who has a history of DRE ≥2 years before enrollment，
4. Participants who has a seizure frequency of ≥2 seizures every month within 3 months before enrollment,
5. Participants and their families are aware of this study and sign informed consent.

Exclusion Criteria:

1. Participants who are in status epilepticus,
2. Participants who are complicated with serious infection, cerebrovascular disease, malignant tumor and other nervous system diseases, with serious dysfunction of heart, liver, kidney and other organs, and with psychiatric disorders,
3. Participants plan invasive therapy, such as operation,
4. Participants who are in pregnancy or lactating,
5. Patients cannot tolerate repeated transcranial magnetic stimulation, or have contraindications of repeated transcranial magnetic stimulation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-28 (Estimated); Primary Completion 2027-03-27 (Estimated); Study Completion 2027-03-27 (Estimated)

PRIMARY OUTCOMES:
seizure reduction rate | Enhanced phase: 2 weeks;Consolidation phase：8 weeks; Maintenance phase：8 weeks; Follow up phase：8 weeks
  A 28-day baseline for seizure frequency will be recorded by the patients themselves or their guardian before therapy and then compare to the frequency after enhanced phase /consolidation/maintenance treatment / 8 weeks after the end of all treatment
responder rate | Enhanced phase: 2 weeks;Consolidation phase：8 weeks; Maintenance phase：8 weeks; Follow up phase：8 weeks
  proportion of people with a 50% or greater reduction in seizure frequency following enhanced phase /consolidation/maintenance treatment / 8 weeks after the end of all treatment

SECONDARY OUTCOMES:
QOLIE-31 scale scores | Enhanced phase: 2 weeks;Consolidation phase：8 weeks; Maintenance phase：8 weeks; Follow up phase：8 weeks
  Quality of Life in Epilepsy-31. Scores range from 0 to 100, with higher scores indicating better quality of life.
scalp electroencephalogram | Enhanced phase: 2 weeks;Consolidation phase：8 weeks; Maintenance phase：8 weeks; Follow up phase：8 weeks
  Routine scalp electroencephalogram at 40 min
MRI | Enhanced phase: 2 weeks;Consolidation phase：8 weeks; Maintenance phase：8 weeks; Follow up phase：8 weeks
  Diffusion tensor imaging，Functional MRI
MoCA | Enhanced phase: 2 weeks;Consolidation phase：8 weeks; Maintenance phase：8 weeks; Follow up phase：8 weeks
  Montreal Cognitive Assessment. A max score is 30 points, and a score ≥ 26 is considered normal.
MMSE | Enhanced phase: 2 weeks;Consolidation phase：8 weeks; Maintenance phase：8 weeks; Follow up phase：8 weeks
  Mini-Mental State Examination. The normal values are defined as: illiterates >17, primary school >20, junior high school or above >24.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No